CLINICAL TRIAL: NCT03503955
Title: Investigation of the Effectiveness of Video Based Games on Upper Extremity Functions in Mild Mental Retardation Diagnosed Cases
Brief Title: Effectiveness of Video Based Games on Upper Extremity Functions in Mild Mental Retardation Diagnosed Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nejla Uzun, Physiotherapist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098
Record Dates: First submitted 2018-04-02; First posted 2018-04-20 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2018-04

CONDITIONS: Mental Retardation; Upper Extremity
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): fine motor skills activities and Leap-Motion virtual reality games
  Interventions: Other: Leap-Motion virtual reality games
- control group (Experimental): fine motor skills activities
  Interventions: Other: fine motor skills activities

INTERVENTIONS:
Other: Leap-Motion virtual reality games — Games that Fizyosoft has prepared on Leap Motion equipment to improve hand and grip activities will be played individually and will focus on running hand, wrist and grip movements
  Arms: study group
Other: fine motor skills activities — activities that stimulate finger movements such as holding, reaching, catching, writing, and strengthening muscles
  Arms: control group

SUMMARY:
With Leap Motion Controller, virtual reality exercises have been implemented more often since 2014, and this technology has benefited more from upper extremity rehabilitation In literature, there are no publications investigating the effectiveness of virtual reality applications on upper extremity functions in cases of mental retardation with Leap Motion.

We think that virtual reality applications with Leap Motion are effective in fine motor skills and grip strength in cases of mental retardation.

The purpose of our work; To Investigation of the Effectiveness of Video Based Games on Upper Extremity Functions in Mild Mental Retardation Diagnosed Cases

DETAILED DESCRIPTION:
For the study group, in addition to fine motor skills activities, 20 min. Leap-Motion virtual reality games, and for the control group only fine motor skill activities will be applied. The study will last 8 weeks, 2 times a week for a total of 16 sessions.The games that Fizyosoft has built on Leap Motion equipment will be played individually and will focus on running hand, wrist and grip movements to improve hand and grip activities of the events. Each game is designed to develop a different hand movement. In this study, CatchaPet and LeapBall of Fizyosoft HandRom products will be used.

"LeapBall," aiming at throwing the ball in the same color as the ball, and Leap Motion sensor games, "CatchaPet," aimed at touching the rabbits out of the holes with repeated wrist flexion / extensional movements, will be preferred by grasping a virtual ball with the fingers of all fingers.

The demographic characteristics of all the cases participating in the study will be recorded.

JEBSON hand function test, Manual Ability Classification System (MACS), 9 Hole Peg Test to measure fine hand skill. JAMAR Hand Dynamometer to measure Hand Grip Force, Pinchmeter to measure finger grip strength. The evaluation will be repeated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* He / she has been diagnosed with mild mental retardation Being between 5 and 18 years of age Ability to adapt to exercises No epileptic epilepsy no cardiac or orthopedic disturbance

Exclusion Criteria:

* Being healthy Not be between 5-18 years

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Jebsen Hand Function Test | Change from Baseline and to the 2 months
  The Jebsen Hand Function Test assesses fine motor skills, weighted and non-weighted hand function activities during performance of activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Ela Tarakcı, Assoc. Prof., Principal Investigator — Istanbul University
Locations (1):
- IstanbulU, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No